CLINICAL TRIAL: NCT04117724
Title: Antibiotic Adherence Practices in Dermatologic Surgery: a Multicenter Prospective Cohort Study
Brief Title: Antibiotic Adherence Practices in Dermatologic Surgery
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833525
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Patients will be asked to complete a 4 question survey assessing adherence. Follow up via patient's preferred method of contact will be conducted after the patient's intended antibiotic completion date and covariates for antibiotic regimens will be recorded including antibiotic type, number of doses, antibiotic duration, reason for non-adherence, pills remaining, and number of other medications.

SUMMARY:
This multi-center prospective observational cohort study will examine the prevalence of non-adherence along with analyze the risk factors of non-adherence for patients presenting to dermatologic surgery. Patients prescribed antibiotics will be invited to participate in the study and appropriate follow up to inquire about antibiotic usage will be conducted. All data will be collected and stored in a secured REDCap database managed by the Penn Dermatologic Surgery Clinical Research Team.

DETAILED DESCRIPTION:
This multi-center prospective observational cohort study will examine the prevalence of non-adherence and analyze the risk factors of non-adherence for patients presenting to dermatologic surgery. Patients prescribed antibiotics will be invited to participate in the study and appropriate follow up to inquire about antibiotic usage will be conducted. Inclusion criteria are 1) Patients with age greater than or equal to 18 who are capable of providing informed consent and 2) Patients who have been prescribed antibiotics following their visit with a dermatologic surgery department. We plan to examine patients who have presented to a dermatologic surgery clinic and were prescribed antibiotics from June 1, 2019 to June 1, 2021 at the University of Pennsylvania Health System and other Institutional Review Board (IRB) approved sites. After obtaining informed consent at their visit to enroll in the study, variables of interest will be collected from patients including name, date of birth (DOB), gender, visit date, contact information, antibiotic regimen, and 4 question survey assessing adherence. Follow up via patient's preferred method of contact will be conducted after the patient's intended antibiotic completion date and covariates for antibiotic regimens will be recorded including antibiotic type, number of doses, antibiotic duration, reason for non-adherence, pills remaining, and number of other medications. All data will be collected and stored in a secured REDCap database managed by the Penn Dermatologic Surgery Clinical Research Team.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than equal to 18
* All patients presenting to one of the dermatologic surgery settings approved by the IRB who are prescribed a post-operative antibiotic regimen

Exclusion Criteria:

* Patients who do not present to or are not prescribed post-operative antibiotics in a dermatologic surgery setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to examine patients who have presented to a dermatologic surgery clinic and were prescribed post-operative antibiotics from June 1, 2019 to June 1, 2021 at the University of Pennsylvania Health System and other IRB approved sites.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of antibiotic non-adherence | Oct 3 2019-July 1 2021
  To analyze the prevalence of antibiotic non-adherence in the dermatologic surgery setting

SECONDARY OUTCOMES:
Risk factors for antibiotic non-adherence | Oct 3 2019-July 1 2021
  To identify risk factors for antibiotic non-adherence

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California, Davis, Davis, California
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Only the study team at the University of Pennsylvania will have access to study data.

REFERENCES:
- [Background] Bae-Harboe YS, Liang CA. Perioperative antibiotic use of dermatologic surgeons in 2012. Dermatol Surg. 2013 Nov;39(11):1592-601. doi: 10.1111/dsu.12272. Epub 2013 Jul 18. PMID 23865410
- [Background] Barbieri JS, Etzkorn JR, Margolis DJ. Use of Antibiotics for Dermatologic Procedures From 2008 to 2016. JAMA Dermatol. 2019 Apr 1;155(4):465-470. doi: 10.1001/jamadermatol.2019.0152. PMID 30825412
- [Background] Kardas P. Patient compliance with antibiotic treatment for respiratory tract infections. J Antimicrob Chemother. 2002 Jun;49(6):897-903. doi: 10.1093/jac/dkf046. PMID 12039881
- [Background] Pechere JC. Parameters important in short antibiotic courses. J Int Med Res. 2000;28 Suppl 1:3A-12A. PMID 11092225
- [Background] Pechere JC. Patients' interviews and misuse of antibiotics. Clin Infect Dis. 2001 Sep 15;33 Suppl 3:S170-3. doi: 10.1086/321844. PMID 11524715
- [Background] Sclar DA, Tartaglione TA, Fine MJ. Overview of issues related to medical compliance with implications for the outpatient management of infectious diseases. Infect Agents Dis. 1994 Oct;3(5):266-73. PMID 7866659